CLINICAL TRIAL: NCT06906718
Title: Evaluation of Long-term Visual Acuity Data After Bilateral Implantation of the Aspheric EDOF Lens ACUNEX® Vario (Model AN6V).
Brief Title: Evaluation of Long-term Visual Acuity Data After Bilateral Implantation of the Aspheric EDOF Lens ACUNEX® Vario
Acronym: ChariteBerAN6V
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teleon Surgical B.V. (Industry)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EA4/120/23
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Intraocular Lens

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AN6V Recipients (Other): Single arm recipients of the IOL
  Interventions: Device: Implantation of an intraocular lens

INTERVENTIONS:
Device: Implantation of an intraocular lens — Successful bilateral IOL implantation into the capsular bag with at least 12 months follow-up.

SUMMARY:
The aim of the ACUNEX® Vario study was to confirm long-term data on the visual quality and contrast sensitivity of an existing EDOF-IOL, which bears the CE mark and has been on the market since 2019.

DETAILED DESCRIPTION:
The monocentric, retro-prospective, uncontrolled clinical study following Art. 82 MDR, §§ 47 MPDG and conducted according ISO 14155 shall confirm the long-term safety and performance of the AN6V - ACUNEX® Vario EDOF-IOL which has been marketed since 2019. This IOL model is designed to provide good distance and intermediate vision.

ELIGIBILITY:
Successful bilateral IOL implantation into the capsular bag with at least 12 months follow-up.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-08-29 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | 12 months
  Visual Acuity at far and intermediate distance.

CONTACTS AND LOCATIONS:
Locations (1):
- Charité University Berlin, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No